CLINICAL TRIAL: NCT07232732
Title: A Phase-1, Parallel-Design, Open-Label, Randomized, Multiple-Dose Escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics of LY3549492 in Healthy Participants With Overweight or Obesity
Brief Title: A Study of LY3549492 in Healthy Participants and Participants With Overweight or Obesity
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27786; J3H-MC-GZNJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3549492 (Treatment Group 1) (Experimental): LY3549492 administered orally.
  Interventions: Drug: LY3549492
- LY3549492 (Treatment Group 2) (Experimental): LY3549492 administered orally.
  Interventions: Drug: LY3549492

INTERVENTIONS:
Drug: LY3549492 — Administered orally

SUMMARY:
The purpose of this study is to see how safe and well-tolerated the drug LY3549492 is and how it behaves in the body, when given in multiple doses to healthy people who are overweight or have obesity. Participation in the study will last approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a hemoglobin A1c level of less than 6.5 percent (%) at screening.
* Have a body mass index (BMI) of 25.0 to 45.0 kilogram per square meter (kg/m²), inclusive, at screening
* Participants assigned male at birth (AMAB) or participants assigned female at birth (AFAB) who are individual of childbearing potential (INOCBP) Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Have obesity induced by endocrine disorders such as Cushing's syndrome or Prader Willi syndrome.
* Have any of the following conditions at screening,

  * supine systolic blood pressure of 160 millimeter of mercury (mmHg) or greater
  * supine diastolic blood pressure of 100 mmHg or greater, or
  * resting pulse rate of greater than 95 beats per minute (bpm) or less than 45 bpm. (Note: white-coat hypertension is excluded; therefore, if a repeated measurement of blood pressure after at least 5 minutes shows values within the range, the participant can be included).
* Have had any of the following within 6-months prior to screening

  * myocardial infarction
  * unstable angina
  * coronary artery bypass graft
  * percutaneous coronary intervention. (Note: diagnostic angiograms are permitted)
  * transient ischemic attack
  * cerebrovascular accident or decompensated congestive heart failure, or
  * New York Health Association Class III or IV heart failure.
* Have serum triglyceride of 5 millimoles per liter (mmol/L) or greater (442 milligrams per deciliter [mg/dL]) at screening
* Have had any exposure to glucagon-like peptide-1 (GLP-1) analogs or other related compounds within the 3 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through end of the Follow-up Period (Week 10)
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3549492 | Predose on Day 1 through end of the Follow-up Period (Week 10)
  PK: Cmax of LY3549492
PK: Observed Drug Trough Concentration (Ctrough) of LY3549492 | Predose on Day 1 through end of the Follow-up Period (Week 10)
  PK: Ctrough of LY3549492
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3549492 | Predose on Day 1 through end of the Follow-up Period (Week 10)
  PK: AUC of LY3549492

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - Fortrea Clinical Research Unit, Dallas, Texas
  - Fortrea Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No